CLINICAL TRIAL: NCT02933268
Title: Determining Feasibility of Randomisation to High vs ad Libitum Water Intake in Polycystic Kidney Disease: The DRINK Randomised Feasibility Trial
Brief Title: High Water Intake in Polycystic Kidney Disease
Acronym: DRINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: PKD Charity (Unknown); Addenbrookes Charitable Trust (Other); British Renal Society & British Kidney Patient Association (Unknown)
Responsible Party: Principal Investigator, Dr Thomas Hiemstra, Honorary Consultant Nephrologist & Senior Trials Research Fellow, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 203565
Record Dates: First submitted 2016-09-18; First posted 2016-10-14 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Autosomal Dominant Polycystic Kidney Disease; Polycystic Kidney Disease; ADPKD; Water; Vasopressin; Dietary
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases; Diabetes Insipidus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ad libitum water intake (Active Comparator): Ad libitum water intake, defined as intake guided by thirst to achieve a target urine osmolality > 300 mOsmo/kg
  Interventions: Other: Ad libitum water intake
- High water intake (Active Comparator): Personalised daily water intake prescription to achieve target urine osmolality < 270 mOsm/kg.
  Interventions: Dietary Supplement: High water intake

INTERVENTIONS:
Dietary Supplement: High water intake — High water intake aimed at achieving an urine osmolality < 270mOsmo/kg. Individualised prescription for each participant based on the free water clearance formula calculation.
  Arms: High water intake
Other: Ad libitum water intake — Water intake guided by thirst
  Arms: Ad libitum water intake

SUMMARY:
DRINK is an open-label randomised controlled feasibility trial of high versus ad libitum water intake in ADPKD.

DETAILED DESCRIPTION:
Autosomal Dominant Polycystic Kidney Disease (PKD) affects 12.5 million people worldwide, and accounts for 7% of those requiring renal replacement therapy. The hormone vasopressin drives cyst growth until ultimately most of the normal functioning kidney tissue is replaced and compressed by cysts over the life course. Half of those affected will require dialysis by the age of 55 years.

Vasopressin blockade has emerged as a viable strategy for altering disease course. High water intake suppresses vasopressin, and may therefore slow cyst growth and consequent disease progression. However, evidence to support high water intake in PKD is lacking, and it is not clear whether patients can adhere sufficiently to a high water intake.

DRINK is a single-centre prospective, open label, parallel group randomised controlled feasibility trial. The primary objective is to establish whether a definitive large randomised trial comparing high versus ad libitum water intake on long-term disease progression is deliverable. Fifty patients will be recruited from the Renal Genetics service at Addenbrooke's Hospital. Participants will be randomly allocated to the high water intake (high) or the ad libitum (standard) water intake group. For the high intake group the aim is to drink large enough volumes of water to achieve and maintain dilute urine (urine osmolality < 270 mOsmo/kg or urine specific gravity ≤ 1.010 ). Multiple methods will be employed to promote adherence these include instruction and education as well as self-monitoring of urine specific gravity twice weekly by participants and the recording of results via a trial specific smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate
* Aged 16 years or older
* Have a diagnosis of ADPKD (fulfilling radiological diagnostic criteria ± genetic evidence)
* eGFR ≥ 20ml/min/1.73m2
* Able to self-monitor urine SG

Exclusion Criteria:

* Inability to provide informed consent
* eGFR < 20ml/min/1.73m2
* Fluid overload states e.g. heart failure, cirrhosis, or requirement for fluid restriction
* Confounding illness impacting on renal disease e.g. concomitant diabetes or glomerulonephritis
* Treatment with diuretics for fluid overload (those on diuretics for hypertension may participate in the trial after a run-in period of 2 weeks)
* Treatment with Tolvaptan in the last 4 weeks
* Pregnancy or breastfeeding

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving a urine osmolality < 270 mOsm/kg | 8 weeks

SECONDARY OUTCOMES:
Urine osmolality | 8 weeks
  Achieved urine osmolality as a surrogate for vasopressin suppression
Proportion of participants that can self-monitor and report urine specific gravity reliably | 8 weeks
Proportion of patients experiencing a serious adverse event | 12 weeks
Acute change in estimated GFR | 4 weeks
  Evaluation of the change form baseline eGFR after 2 weeks
Health-Related Quality of Life (HRQoL) | 12 weeks
  Change from baseline HRQoL as estimated by EQ5D-5L
Recruitment rate | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Himestra, Principal Investigator — Cambridge University Hospital NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] El-Damanawi R, Lee M, Harris T, Mader LB, Bond S, Pavey H, Sandford RN, Wilkinson IB, Burrows A, Woznowski P, Ben-Shlomo Y, Karet Frankl FE, Hiemstra TF. Randomised controlled trial of high versus ad libitum water intake in patients with autosomal dominant polycystic kidney disease: rationale and design of the DRINK feasibility trial. BMJ Open. 2018 May 9;8(5):e022859. doi: 10.1136/bmjopen-2018-022859. PMID 29743334